CLINICAL TRIAL: NCT01866579
Title: Early Retinal Nerve Fiber Layer Change of Ethambutol Optic Neuropathy by Optical Coherence Tomography
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 3-2013-0041
Record Dates: First submitted 2013-05-28; First posted 2013-05-31 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Primary Lung Tuberculosis
Keywords: Retinal Nerve Fiber Layer Thickness, Optical Coherence Tomography, Ethambutol optic neuropathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ethambutol optic neuropathy

SUMMARY:
Ethambutol is widely used as first-line drug, but has serious side effect of optic neuropathy. As previously reported, incidence of ethambutol optic neuropathy is about 1~2%, there was considerable screening efforts and medical cost is increasing. However, there is no effective treatment of ethambutol optic neuropathy or no definite preventable measure. Moreover, multi-drug resistance tuberculosis or extensively drug resistance tuberculosis is emerging, more toxic secondary drug is used in the long-term.

It is known that retinal nerve fiber layer is increased early stage in ethambutol optic neuropathy. So we decide to evaluate the retinal nerve fiber layer thickness measured by optical coherence tomography in longitudinal manner.

ELIGIBILITY:
Inclusion Criteria:

1. Primary lung tuberculosis who has not previously treated
2. Age more than 19 years and less than 70 years old

Exclusion Criteria:

1. spherical equivalent more than +6.00 diopter or less than -6.00 diopter by autorefraction
2. Closed angel or intraocular pressure more than 21 mmHg
3. Best corrected visual acuity less than 0.5 with severe cataract
4. Retinal disorder include branch retinal vein occlusion, diabetic macular edema, wet-type age-related macular degeneration
5. Age less than 20 years or older than 70 years old
6. Any intraocular surgery less than 3 months
7. Intellectual problems or illiterate whom could not obtained informed consent

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who diagnosed with primary lung tuberculosis
Sampling Method: Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2013-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change in Retinal Nerve Fiber Layer thickness measured by optical coherence tomography | Early Retinal Nerve Fiber Layer change of initial before anti-tuberculosis treatment, 4 months after anti-tuberculosis treatment, 6 months after anti-tuberculosis treatmen
  Retinal Nerve Fiber Layer is axon of the retinal ganglion cell. It can be measured by optical coherence tomography. It is non-invasive and good reproducibility method to measure retinal nerve fiber layer in vivo.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, Gangnam Severance Hospital, Seoul, Seoul, South Korea